CLINICAL TRIAL: NCT02189746
Title: A Randomized Trial of Kangaroo Mother Care to Prevent Neonatal Hypothermia - Trials 1A & 1B
Brief Title: Kangaroo Mother Care to Prevent Hypothermia in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Manimaran Ramani, MD, Assistant Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 011
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hypothermia, Newborn
Keywords: Hypothermia; Newborn; Hyperthermia; Kangaroo mother care
MeSH Terms: conditions — Hypothermia; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Continuous Kangaroo Mother Care to 1 hour after birth (Active Comparator): In addition to standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia, the infants will receive continuous KMC most of the time possible from birth to one hour after birth.
  Interventions: Other: Continuous Kangaroo Mother Care to 1 hour after birth
- Standard Kangaroo Mother Care to 1 hour after birth (Sham Comparator): Infants will receive standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia from birth to 1 hour after birth.
  Interventions: Other: Standard Kangaroo Mother Care to 1 hour after birth
- Continuous Kangaroo Mother Care to discharge (Active Comparator): In addition to standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia, the infants will receive continuous KMC most of the time possible from one hour after birth to discharge.
  Interventions: Other: Continuous Kangaroo Mother Care to discharge
- Standard Kangaroo Mother Care to discharge (Sham Comparator): Infants will receive standard WHO thermoregulation care which includes warm delivery rooms, immediate drying, Kangaroo Mother Care (KMC) whenever possible, early and exclusive breastfeeding, postponed bathing and weighing if needed, appropriate bundling and placing the infant in air incubator, radiant heater, or heat mattress if the infant develops hypothermia from 1 hour after birth to discharge.
  Interventions: Other: Standard Kangaroo Mother Care to discharge

INTERVENTIONS:
Other: Continuous Kangaroo Mother Care to 1 hour after birth — Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible until 1 hour of birth. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will be removed from KMC and routine bundling practices will be used. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age.
  Arms: Continuous Kangaroo Mother Care to 1 hour after birth
Other: Standard Kangaroo Mother Care to 1 hour after birth — Infants will receive the standard WHO thermoregulation care of Kangaroo Mother Care for as much as possible until 1 hour of birth, without additional encouragement per study personnel. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. All infants will be resuscitated as usual per Neonatal Resuscitation Program guidelines and hospital standard practices. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will receive standard care which may include removal from KMC and use of routine bundling practices. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age.
  Arms: Standard Kangaroo Mother Care to 1 hour after birth
Other: Continuous Kangaroo Mother Care to discharge — Infants will receive the standard WHO thermoregulation care with encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from one hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), the infant will be removed from KMC and routine bundling practices will be used. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age and again at discharge or 24 hours whichever occurs first.
  Arms: Continuous Kangaroo Mother Care to discharge
Other: Standard Kangaroo Mother Care to discharge — Infants will receive the standard WHO thermoregulation care without additional encouragement from study personnel to keep infant in Kangaroo Mother Care for as much as possible from 1 hour after birth to discharge. In KMC, the naked newborn infant with cap and diaper will be placed prone on mom's bare chest with blanket covering the infant's back. The nursing staff will supervise mother-infant when mother is sleeping with infant in KMC. If infant becomes hyperthermic (>38 degrees Celsius), standard treatment will be given which may include removal from KMC and use of routine bundling practices. The infant's temperature will be taken via axillae with a digital thermometer at one hour of age and again at discharge or 24 hours whichever occurs first.
  Arms: Standard Kangaroo Mother Care to discharge

SUMMARY:
The overall hypothesis is that better adherence to Kangaroo Mother Care (KMC) in combination with existing WHO thermoregulation care will reduce the incidence of moderate hypothermia (32-36 degrees C) or severe hypothermia (<32.0 degrees C) in preterm infants (32-36 6/7 weeks of gestational age) when compared with routine WHO thermoregulation alone.

DETAILED DESCRIPTION:
The overall hypothesis is that better adherence to Kangaroo Mother Care (KMC) in combination with existing World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, KMC whenever possible, early and exclusive breastfeeding, postponement of bathing and weighing, appropriate bundling, and use of air incubator, radiant warmer, or heat mattress if the neonate develops hypothermia) will reduce the incidence of moderate hypothermia (32-36 degrees C) or severe hypothermia (<32.0 degrees C) in preterm infants (32-36 6/7 weeks of gestational age) when compared with routine WHO thermoregulation alone.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age 32-36 6/7 weeks
* Delivery in the hospital

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Minute to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Axillary temperature < 36.0 degrees Celsius | Time of birth to 1 hour
  Temperature taken per axilla for one minute
Axillary Temperature < 36.0 degrees Celsius | At discharge or 24 hours after birth (whichever is first)
  Temperature taken per axilla for one minute

SECONDARY OUTCOMES:
Blood pressure | Duration of hospitalization-expected average of 4 weeks
  Measure of extremity blood pressure per cuff taken during nursery stay.
Blood glucose | Duration of hospitalization-expected average of 4 weeks
  Measure of blood glucose per laboratory value taken per heelstick
Seizure | Duration of hospitalization-expected average of 4 weeks
  Seizure activity diagnosed by medical doctor or nurse. No electroencephalogram will be done.
Respiratory Distress Syndrome (RDS) | Duration of hospitalization-expected average of 4 weeks
  Documentation of increased work of breathing, retractions, and need for oxygen, intubation or surfactant
Sepsis | Duration of hospitalization-expected average of 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis
Neonatal Intensive Care Unit Admission | Duration of hospitalization-expected average of 4 weeks
  Any admission to NICU for need for higher level care
Death | Duration of hospitalization-expected average of 4 weeks
  Cardiorespiratory failure
Any Axillary Temperature < 36.0 degrees Celsius | Duration of hospitalization-expected average of 4 weeks
  Temperature taken per axilla for one minute
Duration of Kangaroo Mother Care | Duration of hospitalization-expected average 4 weeks
  Skin to skin contact between infant and mother

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham; Manimaran Ramani, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia